CLINICAL TRIAL: NCT04596189
Title: Anti-IL4/IL13 Therapy With Dupilumab for Prevention of Refractory Chronic Rhinosinusitis After Endoscopic Sinus Surgery for CRSwNP
Brief Title: Dupilumab for Prevention of Recurrence of CRSwNP After ESS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE20.201
Record Dates: First submitted 2020-10-02; First posted 2020-10-22 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
Keywords: Chronic rhinosinusitis with nasal polyps; Endoscopic sinus surgery; Dupilumab
MeSH Terms: interventions — dupilumab; Mometasone Furoate

STUDY DESIGN:
Intervention Model Description: A placebo-controlled, double blind, prospective, real-world trial in patients with CRSwNP undergoing revision surgery for CRSwNP
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dupilumab (Experimental): Sterile Dupilumab 150 mg/mL will be provided in pre-filled syringes (2.25 total volume) to deliver 300 mg in 2 mL.
  Interventions: Drug: Dupilumab 300 MG in 2 ML Prefilled Syringe; Drug: Mometasone Furoate nasal spray
- Placebo (Placebo Comparator): Sterile placebo for Dupilumab will be provided in identically matching pre-filled syringes to deliver 2 mL.
  Interventions: Other: Placebo; Drug: Mometasone Furoate nasal spray

INTERVENTIONS:
Drug: Dupilumab 300 MG in 2 ML Prefilled Syringe — The Dupilumab will be administered following clinic procedures and blood collection. Patients will be monitored at the study site for at least 30 minutes after injections for signs of hypersensitivity reaction.
  Subcutaneous injection sites should be alternated among the 4 quadrants of the abdomen (avoiding navel and waist areas), the upper thighs or the upper arms, so that the same site is not injected twice consecutively. Injection in the upper arms could be done only by a trained person (caregiver trained by Investigator or Delegate) or health care professional but not the patients themselves.
  Other Names: Dupixent
  Arms: Dupilumab
Other: Placebo — The Placebo will be administered following clinic procedures and blood collection. Patients will be monitored at the study site for at least 30 minutes after injections for signs of hypersensitivity reaction.
  Subcutaneous injection sites should be alternated among the 4 quadrants of the abdomen (avoiding navel and waist areas), the upper thighs or the upper arms, so that the same site is not injected twice consecutively. Injection in the upper arms could be done only by a trained person (caregiver trained by Investigator or Delegate) or health care professional but not the patients themselves.
  Arms: Placebo
Drug: Mometasone Furoate nasal spray — On a daily basis throughout the study, the patient will use a paper diary to record daily use of mometasone furoate nasal spray (MFNS) 50 μg/actuation nasal spray, suspension (refer to the package insert & SmPC for a description, administration details and precautions for use). MFNS is provided in a bottle that contains 18 g (140 actuations) of product formulation. If patient is unable to tolerate 200 micrograms twice a day (total dose 400 micrograms) due to experiencing adverse event, patient may reduce dose to 200 micrograms once per day.
  Other Names: Nasonex

SUMMARY:
The investigators believe that administering Dupilumab during the pre- and peri-operative period of surgery for chronic rhinosinusitis with nasal polyps (CRSwNP) will safely downregulate Type 2 inflammation of the healing sinus environment and will allow for better coordinated and more effective mucosal healing. Specifically, the investigators believe that endoscopic signs and symptoms of recurrence will be reduced in the Dupilumab-treated group, and that this will be reflected in quality of life (QOL). Additionally, by reducing Type 2 inflammation at the time of surgery, Dupilumab may offer an additional benefit by decreasing operative bleeding.

The investigators propose to perform a placebo-controlled, prospective, real-world trial in patients with CRSwNP undergoing revision surgery for CRSwNP to verify whether recurrences after endoscopic sinus surgery (ESS) can be prevented by controlling Type 2 inflammation during the peri-operative period using Dupilumab. A series of seven injections of Dupilumab (or placebo) will be administered to symptomatic patients undergoing ESS for CRSwNP. Beginning 4 weeks prior to surgery and continuing for 8 weeks post-surgery, q2 weekly injections will be administered to reduce Type 2 inflammation at time of ESS and during the post-operative recovery period.

Principal outcome will be absence of recurrence of mucosal oedema of the sinus cavity as assessed by endoscopy. Secondary objectives will assess Polyp size, sinus symptomatology, quality of life, smell and asthma control. Exploratory analyses will assess microbiome and gene expression profiles to better understand molecular mechanisms implicated in CRSwNP pathophysiology, and to identify the pathways implicated by modulation of Type 2 inflammation.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) affects an estimated one in fourteen (7%) Canadians, making it one of the most frequent inflammatory diseases. The human and economic cost of CRS are substantial. Patients affected with chronic sinus disease suffer from headache, facial pain and sinus infections, and experience a reduced quality of life (QOL).The disease has a prolonged course and is frequently resistant to medical therapy.

Current therapeutic strategies involve a combination of nasal irrigations, corticosteroids and antibiotics. Unfortunately, these are rarely curative and raise concerns regarding safety. Oral corticosteroid therapy can lead to severe short and long term adverse effects including diabetes, fractures, psychosis, depression, glaucoma and cataracts. Antibiotic over use is a major driver of development of antibiotic resistance, and antibiotic use in humans in Canada is believed to contribute significantly to this.

In the absence of a response to medical therapy, endoscopic sinus surgery is indicated. Operations for CRS are among the most commonly performed, with over 400 000 surgeries for CRS performed annually in the USA and another 40 000 annually in Canada. However, success is not uniform and a high percentage of patients will continue to manifest signs and symptoms of the disease. Even when managed with a topical intranasal corticosteroid, endoscopic signs of recurrence are observed rapidly after endocopic sinus surgery (ESS) (Stjärne, 2009). In a trial comparing topical mometasone via conventional nasal spray dispenser to placebo, median time to relapse was 173 and 61 days for the mometasone and placebo groups, respectively. This may be improved by use of a more effective form of distribution, such as using budesonide irrigations which improve deposition of steroid in the sinus cavities. In a retrospective analysis of our group limited to a more severely diseased group at higher risk of recurrence, 33% of subjects still showed signs of endoscopic recurrence at 4 month point after surgery (Maniakis, 2014).

Endoscopic sinus surgery may be challenging for patient and surgeon, with risk of complications from trauma to adjacent structures increased by extent of disease and bleeding at time of surgery reducing bleeding. In addition, despite the risks of ESS, recurrence after ESS represents a very important issue as it is rapid and almost ubiquitous.

Patients resistant to surgery generate an individual cost estimated at $10 077/year (Rudmik, 2014). Additional therapeutic options for these patients are currently limited and these patients are currently doomed to continue to suffer despite repeated bouts of antibiotics and surgeries, with patient and society bearing the risks and costs of therapies. Given the frequency, the human and economic burden of refractory CRS, and the deficiencies in effectiveness and adverse effects of current therapies, novel avenues of therapy for CRS are urgently required. Identifying new strategies will require a better understanding of the underlying disease process and identification of new therapeutic targets.

Chronic rhinosinusitis with nasal polyps (CRSwNP) recurrence following surgery is difficult to predict, and the underlying mechanism(s) are not yet well established. However, immune dysfunction with excess Type 2 inflammation, alterations in barrier function and dysbiotic microbiome changes are all believed to play possible roles, which may be targeted by dupilumab. The role of Type 2 inflammation in CRSwNP is well accepted, with the eosinophil described as a characteristic feature of CRSwNP. However, the role of the eosinophil in development of disease has been questioned as a recent trial of a small molecule solution targeting the eosinophil showed effective clearance of eosinophils in polyps, but no effect on symptoms or nasal polyp size. In contrast, Dupilumab, which targets interleukin-4/interleukin-13 (IL4/IL13) cytokines in upstream of IL5, has recently shown in a Phase 3 clinical trial that it reduced symptoms and objective indexes of polyp size and inflammation in CRS. While molecular mechanisms of this remain to be determined, this parallels the effectiveness of other disorders where Type 2 inflammation is central, such as atopic dermatitis and asthma.

How a Type 2 phenotype predisposes to development of sinus disease is unknown but probably represents a multifactorial process. For the past two decades, researchers have postulated that toxic products from degranulation of eosinophilia damaged local structures leading to epithelial breaks and areas of denuded epithelium. The investigators now understand that pro-inflammatory Th2 cytokines are also implicated in epithelial barrier dysfunction. These are not necessarily secreted from the eosinophils, implicating the eosinophil as a downstream marker of the inflammatory process, rather than the primary effector cell. IL4/1L13 has been implicated in epithelial barrier dysfunction. In a series of in-vitro experiments, Wise et al demonstrated that administration of IL4 to an epithelial cell raised in an air-liquid interface, epithelial barrier permeability increased dramatically. Interestingly, this was reversed by anti-IL4. Notable is that this occurred in the absence of eosinophils in the medium, confirming that these effects can occur independently of eosinophil presence.

The epithelial barrier is also believed to play a key role in CRS. Response to tissue injury a key factor in the development of CRS. In CRS, epithelial repair is delayed and dysfunctional. This delayed or inappropriate regeneration of the sinus epithelium and mucosa favours persistence or acquisition of a naltered microbial flora, or microbiome, which then further contributes to the disease process. Firmicutes such as Staphylococcus Aureus and Staphylococcus epidermidis, present in a somewhat mutually exclusive fashion. This new flora may also exacerbate a polarisation of the Type 2 phenotype characteristic of CRSwNP in Caucasians.

It may be possible to interfere with inflammation, epithelial regeneration and repair, and microbiome composition during healing after surgery by modulating Type 2 inflammation. Early rabbit maxillary sinus studies documented formation of polypoid structures in the sinuses following mucosal trauma induced with a cytology brush or following introduction of a respiratory pathogens, with most severe example following simultaneous administration of both. Corticosteroids administered post operatively eliminated polyp formation after injury in this model. However, Type 2-type, eosinophilic polyps only form if the animal has previously been sensitised to develop allergy, suggesting that the Type 2 shift is implicated in the development of nasal polyps. How the Type 2 environment contribute to disease development remains unknown but may either be may directly, via the toxic effect of toxic of eosinophilic granules, or indirectly, by inducing a immunopermissive environment which facilitates bacterial colonisation and persistence. T An understanding of how failures of ESS for CRSwNP develop may be extrapolated form the above experimental findings. Removal of diseased tissue during ESS debrides and removes indwelling inflammatory cells and bacteria and affords an environment which can now be shaped by positive or negative influences. This 'rebirth' concept recently popularized by Bachert et al as the 'reboot' procedure where diseased sinus epithelium is removed surgically to be replaced by 'healthy' cells. However, these new cells regenerate from pluripotential progenitor cells (basal cells, the 'stem cell" of the respiratory mucosa) which may have epigenetic imprinting, or else persistent bacteria may condition to Type 2 environment. By preventing or interfering with these influences during the critical steps of the repair process, the investigators believe they may be able to regenerate a robust epithelium with intact barrier and signaling functions, which attracts normal residential commensals and a "normal" immune status. As all inflammatory and infectious stimulus have been removed, and are not simply lying dormant, it is further theorized that this may produce changes which re-establish normalcy and prevent recurrence of disease. Taken together, the above findings suggest that a Type 2-skewing of the disease process at time of surgery makes surgery more difficult, negatively impacts healing and contributes to the development and persistence of CRS in multiple fashions, marking it as an excellent target for therapeutic intervention.

Managing Type 2 inflammation during the resolution phase is thus an interesting concept which has until now been plagued by practical difficulties. Corticosteroids have historically been the mainstay of therapy for this disease given the frequent presence of Type 2 inflammation and association with asthma. The gold standard of CRSwNP management, a short burst of oral prednisone, has a rapid effect on decrease of polyp size and relief of symptoms but this is of brief duration (≤ 30 days). Additionally, the unfavourable side effect profile precludes long term use.

Novel alternate therapies are urgently required to manage this chronic and debilitating disease. Immunomodulation targeting the Type 2 component of the disease using monoclonal antibodies targeting different aspects of the Type 2 pathway have a potential use in this area, with both anti-IL5 and anti-IL4/IL13 receptors blockers proposed as therapy. The investigators believe that Dupilumab administered during the post-ESS convalescent phase may represent an additional treatment option for CRS.

Population: Thirty-six (36) patients with CRSwNP undergoing a revision surgery for recurrence of CRSwNP, both with and without asthma, will be recruited. Patients will be recruited from the list of patients scheduled for or awaiting surgery, according to usual clinical criteria of obstruction, anosmia, recurrent infections or difficulty with control of asthma. Exclusion criteria include local complications such as mucoceles and tumours, underlying systemic disorders, including sarcoidosis, EGPA (eosinophilic granulomatosis with polyangiitis), Churg-Strauss syndrome, immune deficiency, cystic fibrosis, or a history of neoplasia (excluding basocell carcinoma) within the past two years.

Patients will be homogenous in terms of their symptomatology motivating the operation. In this real-world experience of Dupilumab use, patients will be selected in terms of criteria usually used by clinicians and patients. Polyp size will be required to be at least moderate.

The investigators will ensure homogeneity in patients by:

i) Using standardised, published criteria for definition of patients at high risk of experiencing a recurrence after ESS (Nader ME, 2009).

ii) Using patients at higher risk of failure by restricting study to patients having undergone had at least one prior ESS.

iii) Stipulating a minimal polyp size of at least 2 per side (out of a four point scale) on a Lilleholdt scale.

iv) Rigorous exclusion criteria will exclude polyps secondary to immune deficiency or common pre-existing genetic disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age.
* Patients with bilateral sino-nasal polyposis scheduled for a revision surgery for CRSwNP, according to usual clinical criteria of untolerable obstruction, anosmia, recurrent infections or difficulty with control of asthma.
* Ongoing symptoms (for at least 8 weeks before V1).
* Signed written informed consent.

Exclusion Criteria:

* Patient who has previously been treated with Dupilumab studies
* Patient who has taken:

  * Biologic therapy/systemic immunosuppressant to treat inflammatory disease or autoimmune disease (e.g., rheumatoid arthritis, inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematosus, multiple sclerosis, etc.) within 2 months before V1 or 5 half-lives, whichever is longer.
  * Any experimental mAB within 5 half-lives or within 6 months before V1 if the half-life is unknown.
  * Anti-immunoglobulin E therapy (omalizumab) within 130 days prior to V1.
  * Patients who are receiving leukotriene antagonists/modifiers at V1 unless they are on a continuous treatment for at least 30 days prior to V1.
* Initiation of allergen immunotherapy within 3 months prior to V1 or a plan to begin therapy or change its dose during the run-in period or the randomized treatment period.
* Patients who have undergone any and/or sinus intranasal surgery (including polypectomy) within 6 months before V1.
* Patients who have had a sino-nasal surgery changing the lateral wall structure of the nose making impossible the evaluation of NPS.
* Patients with conditions/concomitant diseases making them non evaluable at V1 or for the primary efficacy endpoint such as:

  * Antrochoanal polyps.
  * Nasal septal deviation that would occlude at least one nostril.
  * Acute sinusitis, nasal infection or upper respiratory infection.
  * Ongoing rhinitis medicamentosa.
* Underlying systemic disorders, including:

  * Cystic fibrosis, allergic granulomatous angiitis (Churg-Strauss syndrome), eosinophilic granulomatosis with polyangiitis (EGPA, Wegener's granulomatosis), Young's syndrome, Kartagener's syndrome or other dyskinetic ciliary syndromes.
* Local complications

  * Radiologic suspicion, or confirmed invasive or expansive fungal rhinosinusitis
  * Mucoceles
* Patients with nasal cavity malignant tumor and benign tumors (eg, papilloma, hemangioma, etc).
* Patients receiving concomitant treatment prohibited in the study.
* Patient is the Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
* Patients meet any contraindications or warning on National Product labeling for MFNS.
* Pregnant or intent to become pregnant during the study, or breast-feeding women.
* Women of childbearing potential (WOCBP) (pre-menopausal female biologically capable of becoming pregnant) who do not fulfill:

  * A confirmed negative serum beta-human chorionic gonadotrophin (β-hCG) test at V1. AND either:
  * An established use of an acceptable contraceptive method: i)Oral, injected, inserted or implanted hormonal contraceptive; ii) Intrauterine device (IUD) with or intrauterine system (IUS) with progestogen; iii) Barrier contraceptive (condom, diaphragm or cervical/vault caps) used with spermicide (foam, gel, film, cream or suppository), if allowed by local regulation. OR,
  * Female sterilization (eg, tubal occlusion, hysterectomy or bilateral salpingectomy).
  * True abstinence in keeping with the preferred and usual lifestyle and if allowed by local regulation; periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) is not an acceptable method of contraception.
  * Postmenopausal women (defined as at least 12 consecutive months with no menses without an alternative medical cause) are not required to use additional contraception.
* Diagnosed active parasitic infection (helminthes); suspected or high risk of parasitic infection, unless clinical and (if necessary) laboratory assessments have ruled out active infection before randomization.
* History of human immunodeficiency virus (HIV) infection or positive HIV screen (Anti HIV-1 and HIV-2 antibodies) at V1.
* A subject with a history of clinically significant renal, hepatic, cardiovascular, metabolic, neurologic, hematologic, ophthalmologic, respiratory, gastrointestinal, cerebrovascular or other significant medical illness or disorder which, in the judgment of the Investigator, could interfere with the study or require treatment that might interfere with the study. Specific examples include but are not limited to uncontrolled diabetes, uncontrolled hypertension, active hepatitis.
* Known or suspected history of immunosuppression, including history of invasive opportunistic infections (eg, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis), despite infection resolution; or unusually frequent, recurrent or prolonged infections, per Investigator's judgment.
* Active tuberculosis, latent untreated tuberculosis or a history of incompletely treated tuberculosis or non-tuberculous mycobacterial infection will be excluded from the study unless it is well documented by a specialist that the patient has been adequately treated and can now start treatment with a biologic agent, in the medical judgment of the Investigator and/or infectious disease specialist. Tuberculosis testing would be performed on a country by country basis according to local guidelines if required by regulatory authorities or ethic committees.
* Evidence of acute or chronic infection requiring treatment with systemic antibacterials, antivirals, antifungals, antiparasitics, or antiprotozoals within 4 weeks before V1 or during the run-in period, or significant viral infections within 4 weeks before V1 that may not have received antiviral treatment.
* Live attenuated vaccinations within 4 weeks prior to Visit 1 or planned live attenuated vaccinations during the study.
* Patients with active autoimmune disease and/or patients using immunosuppressive therapy for autoimmune disease (eg, Hashimoto's thyroiditis, Graves' disease, inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematous, multiple sclerosis, and other neuro-inflammatory disease, psoriasis vulgaris, rheumatoid arthritis), or patients with high titer autoantibodies at V1 who are suspected of having high risk for developing autoimmune disease at the discretion of the Investigator or the Sponsor.
* History of malignancy within 5 years before V1, except completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin.
* Known or suspected alcohol and/or drug abuse.
* Patients with a history of a systemic hypersensitivity reaction, other than localized injection site reaction, to any biologic drug.
* Active hepatitis
* Patients with the following liver injury related criteria at V1:

  * Clinically significant/active underlying hepatobiliary disease. OR,
  * Alanine aminotransferase (ALT) >3 upper limit of normal (ULN).
* Abnormal laboratory values at V1:

  * Creatine phosphokinase (CPK) >10 ULN. OR,
  * Platelets <100 000 cells/mm3. OR,
  * Eosinophils >1500 cells/mm3.
* Conditions/Situations such as: Patients considered by the Investigator or any sub-Investigator as inappropriate for this study for any reason, eg,:

  * Those deemed unable to meet specific protocol requirements, such as scheduled visits.
  * Those deemed unable to administer or tolerate long-term injections as per the patient or the Investigator
  * Presence of any other conditions (eg, geographic, social….) actual or anticipated, that the Investigator feels would restrict or limit the patient's participation for the duration of the study.
* Patient who has withdrawn consent before enrollment/randomization.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with non-recurrence of sinus cavity oedema as assessed endoscopically | Baseline to Week 52
  As it is expected that during the trial period recurrences will remain limited to the confines of the ethmoid sinus cavity and will not extend beyond the middle turbinate, a measuring system capable of capturing oedema as a measure of early changes of polyp formation is required. To this end, a modified version of the Lund-Kennedy grading scale (LK) will be used to assess oedema of the post-ESS sinus cavity.
  Assessment of degree of oedema in patients where nasal polyps do not extend beyond the middle turbinate: 0= No oedema; 1= Mild oedema not obstructing visualisation of surface landmarks or visualisation of the accessory sinus ostia; 2= Oedema obstructing or preventing visualisation of the frontal or sphenoid sinus ostia but not completely filling the sinus cavity; 3= Oedema completely filling the sinus cavity but not extending beyond the middle turbinate.

SECONDARY OUTCOMES:
Percentage of participants with polyp recurrence outside the confines of the sinus cavity(ies) | Baseline to Week 52
  The precentage of patients with nasal polyps extending beyond the confines of the ethmoid cavity of endsoscopy will be recorded.
Percentage of participants requiring a course of oral steroids for recurrence of nasal polyposis. | Baseline to Week 52
  Percent of patients who receive oral steroids for exacerbations of CRSwNP will be compared for the two groups.
Percentage of participants requiring re-operation for recurrence of nasal polyposis | Baseline to Week 52
  Polyp recurrence requiring re-operation will be noted. Polyps extending beyond the middle meatus into the confines of the nasal cavity will be considered as requiring re-operation.
Difference in per-operative bleeding | Week 0 (Day of surgery)
  Difference in per-operative bleeding i) Will be assessed by subjective surgeon evaluation of 'bleeding in the surgical field' during the surgical procedure. Using a standardised grading field, this assesses the surgeon's appraisal of how much bleeding is present during the operation and how much it interferes with visualisation of the associated and underlying structures. This is an important assessment as increased bleeding makes visualisation more difficult and increases the risk of the surgical procedure. (Range=0-3, lower value is better).
  ii) Objective assessment of bleeding. This is performed routinely by tabulating blood loss in the suction apparatus (almost none is lost to other sources such as compresses or gauzes in ESS) while subtracting fluids administered via irrigation and for function of the microdebrider.
Change in total nasal symptomatology | Baseline to Week 52
  Total Nasal Symptom score will be represented on an ordinal scale of 0-9, with lower values indicating less symptoms. Total Nasal Symptom score will be calculated as the sum of the three following symptoms: Nasal obstruction, Nasal secretions, and Facial Pain or Pressure. These symptoms are each individually assessed by questionnaire on a three-point ordinal scale (Range 0-3, lower score is better).
Change in nasal obstruction | Baseline to Week 52
  Change in nasal obstruction will be assessed by questionnaire on a three-point ordinal scale (Range 0-3, lower score is better).
Change in nasal secretions | Baseline to Week 52
  Change in nasal secretions will be assessed by questionnaire on a three-point ordinal scale (Range 0-3, lower score is better).
Change in facial pain | Baseline to Week 52
  Change in facial pain will be assessed by questionnaire on a three-point ordinal scale (Range 0-3, lower score is better).
Change in rhinosinusitis severity visual analog scale (VAS) | Baseline to Week 52
  Change in rhinosinusitis Severity VAS Total nasal symptomatology and burden of sinus conditions will be assessed using a 10 cm visual analogue scale (VAS) (Range 0-10, lower score is better).
Change in Computerized tomography (CT) Scan opacification | Week -4 (4 weeks prior to surgery) to Week 16
  Thin section coronal CT Scan will be obtained at 4 weeks prior to surgery and at 16 weeks post-surgery. These will be graded in a blinded fashion, using the Lund-McKay scoring system. (Range = 0-24, lower value is better).
Change in sense of smell | Baseline to Week 52
  Objective change in sense of smell using the University of Pennsylvania Smell Identification Test with 40 items (UPSIT-40) test. (Range 0-40, higher value is better).
  Subjective change in sense of smell using a three point ordinal scale (''How badly is your sense of smell impaired) .
Change in 22-item Sino-nasal Outcome Test (SNOT-22) | Baseline to Week 52
  Change in quality of life will be assessed using the disease specific 22-item Sino Nasal Outcome Test. Minimally Clinically Important Difference (MCID) score of 8.9 will be used to define i) Response to surgery ii) Deterioration greater than MCID during the post ESS period will be recorded as 'failure'. The total score may range from 0 (no disease) to 110 (worst disease), lower scores representing better health related quality of life.
Change in asthma control | Baseline to Week 52
  Change in asthma control will be assessed using the Asthma Control Questionnaire (ACQ-6) (asthmatic patients only). Range= 0-6, higher score indicated lower asthma control.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Y Desrosiers, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No